CLINICAL TRIAL: NCT02867111
Title: Application of the Sperm Selection Assay in Assisted in Reproductive Technology
Brief Title: Sperm Selection for Infertility Treatment (SSA)
Acronym: SSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Nacional de Córdoba (Other)
Responsible Party: Principal Investigator, Carlos López, MD, Universidad Nacional de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IUMER-1; PIDC2014-0016 (Other Grant/Funding Number: ANPCyT)
Record Dates: First submitted 2016-08-01; First posted 2016-08-15 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Infertility
Keywords: sperm selection; ICSI; Assisted Reproductive Techniques
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- ICSI Control (Other): Intracytoplasmic sperm injection (ICSI), an in vitro fertilization procedure in which a single sperm is injected directly into an egg, with no intervention of the Sperm Selection Assay
  Interventions: Procedure: ICSI
- ICSI + SSA placebo (Placebo Comparator): Intracytoplasmic sperm injection (ICSI), an in vitro fertilization procedure in which a single sperm is injected directly into an egg, with intervention of the Sperm Selection Assay with control solution (culture medium)
  Interventions: Device: Sperm Selection Assay; Procedure: ICSI
- ICSI + SSA Attractant substance (Experimental): Intracytoplasmic sperm injection (ICSI), an in vitro fertilization procedure in which a single sperm is injected directly into an egg, with intervention of the Sperm Selection Assay with attractant solution (attractant diluted in culture medium at 10 pM)
  Interventions: Device: Sperm Selection Assay; Other: Attractant Substance; Procedure: ICSI

INTERVENTIONS:
Device: Sperm Selection Assay — Sperm Selection Assay (SSA) that allow the investigators to select functional spermatozoa, which are capacitated, with intact DNA, reduced oxidative stress and with good viability and motility, on the basis of sperm chemotaxis towards a physiological attractant molecule.
  Other Names: SSA
  Arms: ICSI + SSA Attractant substance; ICSI + SSA placebo
Other: Attractant Substance — Capacitated spermatozoa may be oriented by following an increasing concentration gradient of an attractant molecule, a phenomenon called sperm chemotaxis. This is a guidance mechanism observed in vitro, which may transport and retain spermatozoa at the fertilization site. Though several molecules have been suggested to attract human spermatozoa, in the context of gamete interaction prior to fertilization, progesterone has biological importance for several reasons. After ovulation, this hormone is secreted by the cumulus cells that surround the oocyte, diffusing to form a molecular gradient toward the periphery of the cumulus and beyond. Notably, a gradient of very low concentrations (picomolar) of progesterone is sufficient to chemically attract capacitated human spermatozoa
  Arms: ICSI + SSA Attractant substance
Procedure: ICSI — An in vitro fertilization procedure in which a single sperm is injected directly into an egg
  Other Names: Intracytoplasmatic Sperm Injection

SUMMARY:
Infertility is considered a disease by the World Health Organization and it is increasing worldwide affecting more than 70 million couples. About 50% of the cases are due to male inability to fertilize the oocyte. In the last 40 years, several techniques, known as Assisted Reproduction Technology (ART) have been developed to treat infertility, but the efficiency is still relatively low (around 30%) whereas the remaining 70% attempts again several times, an expensive and emotionally moving treatment. Over 4million of infertility treatments are practiced around the world per year and a 50% increment is expected over the next 6years. Even though ART allows the birth of babies that would be impossible under natural circumstances, it is still necessary to improve the procedures in order to increase treatment efficiency. The success of ART depends, to some extent, on sperm quality. Indeed, the relevance of spermatozoa quality is notorious even beyond fertilization, extending to embryo development and implantation. In this context, it has been developed a new technology that allows the selection of those spermatozoa at their best functional state (Sperm Selection Assay, SSA; Patent approved for USA and Europe, pending for Japan and Argentina). This method is based on the attraction of spermatozoa ready to fertilize the egg, towards a physiological attractant molecule. The SSA may be applied to improve diagnosis and infertility treatment. The investigators hypothesis states that the use of the SSA will improve the number of good-quality embryos which are the ones to be transferred by intracytoplasmic sperm injection (ICSI), providing a healthy embryo development. The protocol involves three experimental groups where the SSA will be used or not, before performing the ICSI: 1)SSA containing the sperm attractant molecule, 2)SSA without the attractant molecule, and 3)without SSA. The patient inclusion criteria involve female factors associated to tubal obstruction and/or endometriosis and male factors associated to sperm disability. Several outcome parameters will be determined, the percentage of fertilization, embryo quality, rate of pregnancy and rate of birth. The study will be carried out in the Universitarian Institute of Reproductive Medicine (IUMER) which has been recently established in a public hospital depending on the National University of Córdoba, offering free high complexity infertility treatment to patients without health insurance or economic support

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis for primary and secondary infertility
* Healthy females or females with tubal obstruction (uni or bilateral) and/or endometriosis.
* Clinical diagnosis for unexplained infertility.
* Females between 18 and 40 years old.
* Healthy males between 18 and 50 years old.
* Males with oligozoospermia, teratozoospermia, asthenozoospermia or asthenoteratozoospermia.

Exclusion Criteria:

* Low complexity assisted reproductive techniques
* In vitro fertilization treatment
* Other medical diagnosis of female infertility besides the inclusion criteria
* Males with oligoasthenoteratozoospermia and oligoasthenozoospermia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Fertilization rate | within 24 hs
  Fertilization rate= number of fertilized oocyte (oocytes with 2 pronuclei) / Total of injected oocytes in metaphase II

SECONDARY OUTCOMES:
Embryo quality | within 48 to 66hs post injection
  Grade I: Embryos with blastomeres of same size without fragmentation (degree 1) with clear and homogeneous cytoplasm, II: Embryos with blastomeres of the same size and less than 30% of fragmentation (degree 2 or 3), III: Embryos with blastomeres of different size and 0% of fragmentation (degree 1), IV: Embryos with blastomeres of the same or different sizes with 30 to 50% of fragmentation (degree 4), V: Embryos with more than 50% of fragmentation (degree 5).
Transferable embryo rate | within 72hs post injection
  Transferable embryo rate= Number of embryos in condition to be transferred / Number of oocytes
Pregnancy rate | within 30 days post injection
  pregnancy rate= Number of positive implantation / Total of patients with transferred embryos
Birth rate | Up to 42 weeks after positive implantation
  Birth rate= Number or live birth / Total of positive pregnancy
Implantation yield | 72 hs post injection
  Implantation rate= Number of implanted embryos / Number of transferred embryos
Division rate | within 24-72 hs post injection
  Division rate= divided embryos / oocytes with 2 pronuclei
Fecundation failures in ICSI rate | Within every cycle of ICSI
  ICSI cycles with no oocyte fecundated / ICSI cycles
Blastocyst formation rate | within 3 to 5 days after injection
  number of embryos that reach blastocyst stage / number of total embryos
Abortion rate | within 3 months post injection
  number of abortions / number of pregnancies
multiple embryo rate | within a month post injection
  number of embryos with more than one gestational sac / total of embryos
clinic gestational rate | within one month after injection
  number of cycles when gestational sac is observed / total of cycles
biochemist gestational rate | within 45 days after injection
  number of cycles with positive beta human chorionic gonadotropin without gestational sac / total of cycles
Cycles without transferred embryos rate | within 2 months after recruitment
  number of cycles without transfer / number of cycles with ovaric puncture
Degree Fragmentation | within 48hs to 66hs post injection
  the embryos will be classified according with the size and distribution of cytoplasmic fragments in 5 categories. 1- Without fragments, 2- Up to 10% of fragmentation, 3- Up to 30% of fragmentation, 4- Between 30 to 50% of fragmentation and 5- More than 50% of fragmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Laura C. Giojalas, PhD, Principal Investigator — National University of Cordoba
Locations (2):
- Argentina (2):
  - HALITUS Instituto Médico, Buenos Aires, Buenos Aires F.D.
  - Instituto Universitario de Medicina Reproductiva (IUMER), Córdoba, Córdoba Province

IPD SHARING:
Plan to Share IPD: No